CLINICAL TRIAL: NCT02203760
Title: Pazopanib Vs. Pazopanib Plus Gemcitabine in Patients with Relapsed or Metastatic Uterine Leiomyosarcomas or Uterine Carcinosarcomas: a Multi-center, Randomized Phase-II Clinical Trial of the NOGGO and AGO - PazoDoble -
Brief Title: Pazopanib Vs. Pazopanib Plus Gemcitabine
Acronym: PazoDoble
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Collaborators: Novartis Pharmaceuticals (Industry); medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOGGO U1; 2012-003810-15 (EudraCT Number)
Record Dates: First submitted 2014-05-05; First posted 2014-07-30 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Leiomyosarcoma or Carcinosarcoma
Keywords: Relapsed/metastatic uterine leiomyosarcomas/carcinosarcomas
MeSH Terms: conditions — Leiomyosarcoma; Carcinosarcoma; Recurrence | interventions — pazopanib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pazopanib plus Gemcitabine (Experimental): Arm A: Pazopanib 800 mg orally once daily plus Gemcitabine 1000 mg/m2 i.v. over 30 min d 1 and d 8 q3w or
  Interventions: Drug: Pazopanib plus Gemcitabine
- Pazopanib (Active Comparator): Pazopanib 800 mg orally once daily
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib plus Gemcitabine — Pazopanib 800 mg orally once daily plus Gemcitabine 1000 mg/m2 i.v. over 30 min d 1 and d 8 q3w or
  Other Names: Votrient and Gemzar
  Arms: Pazopanib plus Gemcitabine
Drug: Pazopanib — Pazopanib 800 mg orally once daily
  Other Names: Votrient
  Arms: Pazopanib

SUMMARY:
This study is a prospective, randomized, open-label, multicenter phase II trial in order to determine progression-free survival of patients with refractory or relapsed metastatic uterine leiomyosarcomas or other metastatic uterine tumours.

DETAILED DESCRIPTION:
Study design:

This study is a prospective, randomized, open-label, multicenter phase II trial in order to determine progression-free survival of patients with refractory or relapsed metastatic uterine leiomyosarcomas or other metastatic uterine tumours.

Indication:

Relapsed or metastatic uterine leiomyosarcomas or carcinosarcomas

Randomization:

Patients with uterine leiomyosarcomas will be randomized in a 1:1-fashion to receive the following therapy

* Arm A: Pazopanib 800 mg orally once daily plus Gemcitabine 1000 mg/m2 i.v. over 30 min d 1 and d 8 q3w or
* Arm B: Pazopanib 800 mg orally once daily Patients with uterine carcinosarcomas will be treated according to Arm A.

Planned number of patients:

87 patients with uterine leiomyosarcomas 20 patients with uterine carcinosarcomas

Treatment schedules:

Patients with uterine leiomyosarcomas will be randomized in a 1:1-fashion to receive the following therapy • Arm A (experimental arm / combination arm): Pazopanib 800 mg orally once daily plus Gemcitabine 1000 mg/m2 i.v. over 30 min d 1 and d 8 q3w or

• Arm B (control arm / monotherapy arm): Pazopanib 800 mg orally once daily Patients with uterine carcinosarcomas will be treated according to Arm A.

Planned treatment duration per subject:

Patients continue on study treatment until disease progression, death, unacceptable toxicity or withdrawal of consent for any reason.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up. Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol
2. Histologically or cytological confirmed uterine leiomyosarcoma or uterine carcinosarcoma including any subtypes
3. Patients with a contraindication for doxorubicin OR patients must have received prior chemotherapies
4. For patients with prior anthracycline therapy normal cardiac function with LVEF at least 50% must be assessed by quantitative echocardiogram or MUGA scan
5. Prior Gemcitabine containing chemotherapy is permitted provided that at least 8 weeks have elapsed since the last dose of therapy
6. ECOG performance status 0-1
7. At least 18 years old
8. Measurable disease according to RECIST v 1.1 criteria (in case of tumour debulking - staging CT-scan after surgery)
9. Able to swallow and retain oral medication
10. Adequate organ system function as defined in Table 1

Table 1: Definitions for Adequate Organ Function System Laboratory Values Hematologic Absolute neutrophil count (ANC) > = 1.5 X 109/L Hemoglobin1 > = 9 g/dL (5.6 mmol/L) Platelets > = 100 X 109/L Prothrombin time (PT) or international normalized ratio (INR)4 <= 1.2 X upper limit of normal (ULN) Partial thromboplastin time (PTT) <=1.2 X ULN Hepatic2 Total bilirubin <= 1.5 X ULN AST and ALT <= 2.5 X ULN Renal Serum creatinine <= 1.5 mg/dL (133 µmol/L)

Or, if greater than 1.5 mg/dL:

Calculated creatinine clearance > = 50 mL/min

Urine Protein to Creatinine Ratio (UPC)3 < 1

1. Subjects may not have had a transfusion within 7 days prior to screening assessment.
2. Concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN are not permitted
3. If UPC > = 1, then a 24-hour urine protein must be assessed. Subjects must have a 24-hour urine protein value <1g to be eligible.
4. Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation

11. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:

* A hysterectomy
* A bilateral oophorectomy (ovariectomy)
* A bilateral tubal ligation
* Is post-menopausal Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥ 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value >40 mIU/mL and an estradiol value < 40pg/mL (<140 pmol/L).

Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT

OR

Negative serum pregnancy test of women of childbearing potential performed within 1 week prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. Acceptable contraceptive methods, when used consistently and in accordance with the product label and the instructions of the physicians are as followed for 14 days before exposure to investigational product, through the dosing period and for at least 21 days after the last dose of investigational product:

* Complete abstinence from sexual intercourse
* Oral contraceptive, either combined or progestogen alone
* Injectable progestogen
* Implants of levonorgestrel
* Estrogenic vaginal ring
* Percutaneous contraceptive patches
* Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
* Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
* Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository) Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

Exclusion Criteria:

1. Prior malignancy

   • Note: Subjects who have had another malignancy and have been disease-free for 5 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
2. Patient has received prior treatment with any anti-angiogenic agent including bevacizumab and tyrosine kinase inhibitors
3. Active malignancy or any malignancy in the last 5 years prior to first dose of study drug other than LMS and CS
4. History or clinical evidence of central nervous system (CNS) or leptomeningeal metastases, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug. Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases
5. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

   * Active peptic ulcer disease
   * Known intraluminal metastatic lesion/s with risk of bleeding
   * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
   * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment
   * Grade 3/4 diarrhea
6. Corrected QT interval (QTc) > 450 Milliseconds using Barzett's formula
7. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Cardiac angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Coronary artery bypass graft surgery
   * Symptomatic peripheral vascular disease
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
   * Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90 mmHg].

   Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. BP must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP / DBP values from each BP assessment must be <140/90 mmHg in order for a subject to be eligible for the study (refer to study protocol for details on BP control and re-assessment prior to study enrollment)
8. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

   • Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
9. Major surgery or trauma within 28 days prior to study enrolment or any non- healing wound, fracture or ulcer (procedures such as catheter placement not considered to be major)
10. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to Pazopanib or Gemcitabine
11. Evidence of active bleeding or bleeding diathesis
12. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
13. Hemoptysis in excess of 2.5 mL(or one half teaspoon) within 8 weeks prior to the first dose of study drug
14. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
15. Unable or unwilling to discontinue use of prohibited medications listed in the study protocol for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study
16. Treatment with any of the following anti-cancer therapies

    * Radiation therapy, surgery or tumour embolization within 14 days prior to the first dose of study drug
    * Chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug
17. Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia
18. Pregnancy (for women of childbearing potential to be confirmed by negative serum pregnancy test) or lactation period

    Women of childbearing potential:

    missing contraception (Pearl-Index <1, e.g. hormonal contraception including the combined oral contraceptive pill, the transdermal patch, and the contraceptive vaginal ring, intrauterine devices or sterilization) for 14 days before exposure to investigational product, during study treatment and for at least 21 days after the last dose of investigational product.
19. Medical or psychological conditions that would not permit the subject to complete the study or sign informed consent
20. Legal incapacity or limited legal capacity
21. Participation in another clinical study with experimental therapy within 30 days prior to study enrolment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival assessed as rate of patients without progression Second malignancy or clinical progression - patients with unknown or missing PFS will be treated as non-responder | 6 months

SECONDARY OUTCOMES:
Objective response rate (RECIST v1.1 criteria) | One year
  Time to progression (TTP) of a patient being defined as the time in months from start of the first therapy cycle until PD is observed
Objective response rate (RECIST v1.1 criteria) | One year
  Overall survival (OS) calculated from the day of study enrolment until the day of death
Objective response rate (RECIST v1.1 criteria) | one year
  Progression-free survival (PFS) calculated from the day of study enrolment until the day of progression/death
Safety - side effects | One year
  Toxicity and tolerability
Quality of life (EORTC QLQ-C30) | One year
  Quality of life (EORTC QLQ-C30)
Translational research program | One year
  Translational research within a tumour bank

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Mustea, Prof. Dr. med., Study Chair — University Hospital, Bonn
Locations (9):
- Germany (9):
  - Universitätsklinikum Bonn, Bonn, Bonn
  - Helios Klinikum Berlin-Buch, Klinik für Onkologie und Paliativmedizin, Berlin, Germany
  - Universitätsmedizin Greifswald Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, Greifswald, Greifswald
  - Helios Klinikum Bad Saarow, Hämatologie, Onkologie und Palliativmedizin, Sarkomzentrum, Bad Saarow
  - Universitätsmedizin Berlin Charité Campus Virchow-Klinikum, Berlin
  - Universitätsklinik Carl Gustav Carus der Technischen Universität Dresden Klinik für Frauenheilkunde und Geburtshilfe, Dresden
  - Kliniken-Essen-Mitte Evang. Huyssens-Stiftung Klinik für Senologie / Brustzentrum, Essen
  - Universitätsklinikum Jena, Jena
  - Universitätsfrauenklinik Tübingen, Tübingen